CLINICAL TRIAL: NCT00237601
Title: Home or Home-like Hospital Birth for Low-risk Nulliparae: Does it Matter?
Brief Title: Home or Home-like Hospital Birth
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Collaborators: School for Midwifery Maastricht (Unknown)
Responsible Party: Jan G. Nijhuis, Prof MD PhD, Maastricht University Medical Centre
Other Study IDs: PF 198
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Last update posted 2010-04-02 (Estimated); Status verified 2010-04

CONDITIONS: Pregnancy
Keywords: Home birth; Hospital birth; Midwifery; Effectivity; Efficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Women with the intention to give birth at home
  Interventions: Other: obstetric care
- 2: Women with the intention to give birth in a short-stay hospital setting
  Interventions: Other: obstetric care

INTERVENTIONS:
Other: obstetric care

SUMMARY:
In the Netherlands, which has about 200.000 births per year, maternity care is provided by midwives or general practitioners unless medical reasons necessitate specialist obstetric care. Women with low risk pregnancies are free to decide where to give birth, attended by their midwife or general practitioner, at home or in the hospital, from which they are then discharged within 24 hours. In the Netherlands these hospital births are referred to as "poliklinische bevallingen" (i.e. outpatient deliveries) to indicate that they do not involve formal hospitalisation, or as "verplaatste thuisbevalling" (i.e. relocated home births) to indicate that they are supervised by the same caregivers as the home births without involvement of specialist obstetricians.

In the last two decades a marked increase in the referral rate to obstetricians during childbirth has occurred, especially for nulliparae, both in planned home births and planned hospital births (outpatient deliveries). 90% from all primigravidae will start their pregnancy under care of the primary caregiver (midwife of general practitioner). During the pregnancy 30% will be referred to the secondary caregiver (obstetrician specialist). The other 60% will start labor guided by the primary caregiver. More than 50% of these women will be referred to the obstetrician during labor.

Despite this unique situation of the Dutch maternity care, the differences between home and hospital birth (outpatient deliveries) with regard to effectivity and efficiency have never been investigated. It is also unclear if pregnant women are informed about a 50% risk of being transported to the secondary caregiver/ hospital during labor at home. Neither do we know what their experiences are.

This study aims to investigate the differences between home and hospital deliveries under care of the primary caregiver with regard to effectivity (costs) and efficiency (patient satisfaction) of care.

ELIGIBILITY:
Inclusion Criteria:

* Primiparae
* No medical indication for specialistic care
* The pregnant woman will be able to give birth at home or at a hospital
* The woman and her partner will be fluent in the Dutch language

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Women with a low-risk pregnancy under the care of an independent midwife. Women are free to choose where to give birth, at home or in a short-stay hospital setting. The women are fluent in de Dutch language.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2006-01; Primary Completion 2008-03 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
primary outcome: referral rate to secondary care, preferences of women and partners with regard to place of birth. Secondary outcome: costs of home birth and hospital births satisfaction of obstetric care

CONTACTS AND LOCATIONS:
Overall Officials: Jan G. Nijhuis, Prof dr MD PhD, Study Chair — Maastricht University Medical Center; Marijke JC Hendrix, MBA, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Academic Hospital Maastricht, Maastricht, Netherlands

REFERENCES:
- [Derived] Aldana-Bitar J, Moore J, Manubolu VS, Dahal S, Verghese D, Lakshmanan S, Hussein L, Crabtree T, Jonas R, Min JK, Earls JP, Budoff MJ. Plaque Progression Differences Between Apixaban and Rivaroxaban in Patients With Atrial Fibrillation Measured With Cardiac Computed Tomography and Plaque Quantification. Am J Ther. 2023 Jul-Aug 01;30(4):e313-e320. doi: 10.1097/MJT.0000000000001569. Epub 2022 Oct 18. PMID 36731003